CLINICAL TRIAL: NCT02986451
Title: Efficacy and Safety Study of BiRD (Biaxin [Clarithromycin]/Revlimid [Lenalidomide]/Dexamethasone) Combination Therapy in Relapsed/Refractory Myeloma
Brief Title: Clarithromycin,Lenalidomide and Dexamethasone for Relapsed/Refractory Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: China Food and Drug Administration (Other Government)
Responsible Party: Principal Investigator, wanghua, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-2016
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Relapse/Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Clarithromycin; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): All patients received clarithromycin, lenalidomide, and dexamethasone in 28-day cycles. Dexamethasone (40 mg) was given orally on days 1, 8, 15, and 22. Clarithromycin (500 mg) was given orally twice daily.Lenalidomide (25 mg) was given orally daily on days 1 to 21
  Interventions: Drug: clarithromycin; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: clarithromycin — Clarithromycin 500mg PO twice daily on days 1-28 for a 28-day cycle.
  Other Names: Biaxin
Drug: Lenalidomide — Lenalidomide 25mg PO daily on days 1-21 of a 28-day cycle
  Other Names: Revlimid
Drug: Dexamethasone — Dexamethasone 40mg PO will be given on days 1, 8, 15, 22 of a 28-day cycle.
  Other Names: hexadecadrol

SUMMARY:
This phase II study investigating the efficacy and safety of a combination of biaxin,lenalidomide and dexamethasone in subjects with relapsed/refractory MM.

DETAILED DESCRIPTION:
The combination of lenalidomide and dexamethasone is effective in increasing the response rate, time to progression, and overall survival in patients with relapsed or refractory myeloma.Clarithromycin is an antibiotic that has shown efficacy in association with steroids and lenalidomide.Clarithromycin, lenalidomide and dexamethasone (BiRd) in newly diagnosed MM has yielded an overall response rates (ORR) of 93% and a progression-free survival (PFS) of 43 months.No prospective study of BiRd to treat relapsed or refractory myeloma has been reported so far.The goal of this phase 2 clinical trial was to assess the response rate and toxicity of a combination regimen of clarithromycin (Biaxin), lenalidomide (Revlimid), and dexamethasone (BiRD) for the treatment of relapsed/refractory MM.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a previous diagnosis of multiple myeloma
* Patient requires retreatment for multiple myeloma
* Subject has measurable disease as defined by > 0.5 g/dL serum monoclonal protein, >10 mg/dL involved serum free light chain (either kappa or lambda) provided that the serum free light chain ratio is abnormal, >0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s) of at least 1cm in greatest dimension as measured by either CT scanning or MRI
* Subject has a Karnofsky performance status ≥60% (>50% if due to bony involvement of myeloma (see Appendix IV)
* Subject has a life expectancy ≥ 3 months
* Subjects must meet the following laboratory parameters:

Absolute neutrophil count (ANC) ≥750 cells/mm3 (1.0 x 109/L) Hemoglobin ≥ 7 g/dL Platelet count ≥ 75,000/mm3 (30 x 109/L if extensive bone marrow infiltration) Serum SGOT/AST <3.0 x upper limits of normal (ULN) Serum SGPT/ALT <3.0 x upper limits of normal (ULN) Serum total bilirubin <2.0 mg/dL (34 µmol/L) Creatinine clearance ≥ 30 cc/min

Exclusion Criteria:

* Subject has immeasurable MM (no measurable monoclonal protein, free light chains in blood or urine, or measureable plasmacytoma on radiologic scanning)
* Subject has a prior history of other malignancies unless disease-free for ≥ 5 years, except for basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or localized prostate cancer with Gleason score < 7 with stable prostate specific antigen (PSA) levels
* Subject has had myocardial infarction within 6 months prior to enrollment, or NYHA (New York Hospital Association) Class III or IV heart failure (see Appendix VI), Ejection Fraction < 35%, uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Female subject who is pregnant or lactating
* Subject has known HIV infection
* Subject has known active hepatitis B or hepatitis C infection
* Subject has active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program
* Subject is unable to reliably take oral medications
* Subject has known hypersensitivity to dexamethasone,cyclophosphamide,paclitaxel
* Subject has a history of thromboembolic event within the past 4 weeks prior to enrollment
* Subject has any clinically significant medical or psychiatric disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 30 months
  ORR is defined as the proportion of patients with CR, nCR or partial response (PR) based on modified EBMT criteria per investigator assessment

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 30 months
  PFS, defined as time from first dose of study treatment to progression or death due to any cause, as assessed by investigator
Overall survival (OS) | 30 months
  OS, defined as time from first dose of study treatment to death
Safety of combination therapy assessed using the National Cancer institute-Common Toxicology Criteria (NCI-CTC) grade scale for AEs and Lab assessments | 30 months
  Safety of combination therapy (Clarithromycin,lenalidomide and dexamethasone) as assessed by toxicity, which will be assessed using the National Cancer Institute-Common Toxicology Criteria (NCI-CTC) grading scale for Adverse Events and for laboratory assessments (v4.03) that include biochemistry, hematology, urinalysis; special safety assessments that include LVEF, Thyroid function Creatinine clearance and ECGs (electrocardiograms).
Genomic Predictors of Response Rate and PFS | 30 months
  Blood (about 1-2 tablespoons) collected for biomarker and routine tests and to evaluate the ORR and PFS.

CONTACTS AND LOCATIONS:
Overall Officials: zhongjun xia, MD., Principal Investigator — hematological oncology department
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No